CLINICAL TRIAL: NCT01352390
Title: The Effect of a Coloring Prompt on Health Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 813606
Record Dates: First submitted 2011-05-06; First posted 2011-05-11 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: In Need of a Pap Smear (Cervical Cancer Screening); In Need of a Blood Pressure Check (Hypertension Screening); In Need of a Cholesterol Test (Lipid Disorder Screening); In Need of a Fasting Plasma Glucose Test (Diabetes)
Keywords: behavioral economics; nudge; artwork; Pap smear; Blood pressure check; Cholesterol test; Fasting plasma glucose test
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Condition (Active Comparator): A basic reminder mailing will prompt each subject to receive a health test as specified on the mailing
  Interventions: Behavioral: Control Condition
- Artwork Prompt Condition (Experimental): A basic reminder mailing will prompt each subject to give their child a reminder postcard to color
  Interventions: Behavioral: Planning Prompt

INTERVENTIONS:
Behavioral: Planning Prompt — A prompt to have their child their health test reminder mailing to color
  Arms: Artwork Prompt Condition
Behavioral: Control Condition — A basic reminder mailing will prompt each subject to get a health test as specified on the mailing
  Arms: Control Condition

SUMMARY:
The goal of this project is to determine whether prompting the recipient of a health reminder mailing to ask his or her 4-9 year-old child to color on the reminder could increase engagement with the targeted health behavior

DETAILED DESCRIPTION:
The investigators will randomly assign some individuals with 4-9 year old children to receive colorful reminders to engage in a given health behavior. Others will receive identical reminders along with a prompt to share the reminder sheet with their child so it can be turned into a piece of art. The investigators are interested in whether the coloring prompt will lead the reminder to stay in the home for longer, be placed on the refrigerator, etc. and thus result in an increase in compliance with the recommended health behavior.

ELIGIBILITY:
Inclusion Criteria:

* Indications according to Spring 2011 CDC criteria for a Pap smear
* Indications according to Spring 2011 CDC criteria for a blood pressure check
* Indications according to Spring 2011 CDC criteria for a cholesterol test
* Indications according to Spring 2011 CDC criteria for a fasting plasma glucose test
* Employee at partner corporation that implemented the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8711 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants that schedule an appointment for receipt of a Pap smear. | up to 52 weeks

SECONDARY OUTCOMES:
Number of Participants that schedule an appointment for receipt of a Blood pressure check | up to 52 weeks
Number of Participants that schedule an appointment for receipt of a Cholesterol test | up to 52 weeks
Number of Participants that schedule an appointment for receipt of a Fasting plasma glucose test | up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States